CLINICAL TRIAL: NCT05520203
Title: Role Development, Implementation and Evaluation of Nurse Practitioners in a Belgian University Hospital.
Brief Title: Role Development, Implementation and Evaluation of Nurse Practitioners
Acronym: NUPRA
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: KW2196/DVE/001/001; B6702021000685 (Other: Ethics Committee UZ Gent); B6702021000300 (Other: Ethics Committee UZ Gent); B6702021000479 (Other: Ethics Committee UZ Gent); B6702021000046 (Other: Ethics Committee UZ Gent)
Record Dates: First submitted 2022-04-15; First posted 2022-08-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Nurse Practitioners; Implementation Research; Quality of Care
Keywords: advanced practice nursing; interdisciplinary health team; participatory action research; longitudinal mixed methods study; nursing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Patient - cohort 1: Patients (and their parents) recruited before introduction of the NP
  Interventions: Other: Care provided by the Nurse Practitioner
- Patient - cohort 2: Patients (and their parents) recruited after introduction of the NP
  Interventions: Other: Care provided by the Nurse Practitioner
- Healthcare providers: Healthcare providers involved in the process of development, implementation and evaluation as well as all healthcare providers who come into close contact with the Nurse Practitioner
  Interventions: Other: Care provided by the Nurse Practitioner

INTERVENTIONS:
Other: Care provided by the Nurse Practitioner — Introduction of a Nurse Practitioner in the interdisciplinary care team

SUMMARY:
Hospitals face new challenges in providing sustainable high quality care as the prevalence of chronic conditions, multimorbidity and the complexity of care increases. The high burden on healthcare teams, the growing costs and the increasing scarcity in healthcare providers (HCPs) result in unmet needs of patients and their families and a high workload on HCPs. Worldwide there is growing recognition that new care models integrating nurse practitioners (NPs) in interdisciplinary teams could contribute to respond to these challenges.

ANP is defined as an "advanced practice nurse (APN) who integrates clinical skills associated with nursing and medicine in order to assess, diagnose and manage patients in primary healthcare settings and acute care populations as well as ongoing care for populations with chronic illness".

Despite the proven benefits of integrating NPs in interdisciplinary teams, the introduction of NPs in Belgium is at an early stage. Advanced practice nurses, including NPs, are formally recognized in Belgium since 2019, but there is still no legal framework in which additional rights or agreements compared to other nursing groups are defined. Given the early stage of introduction, little is known about the development, implementation and impact of NPs in the Belgian health care context. Insights in implementation processes and the effectiveness of NP roles at different levels can inform healthcare managers and policy makers for future (nation-wide) implementation in a hospital setting.

The overall objective of this longitudinal pre-post mixed methods study is to develop, implement and evaluate the integration of the role of NPs in four different departments in a Belgian university hospital.

DETAILED DESCRIPTION:
A mixed methods design is used to enrich the gathered data, resulting in an integrated approach for addressing the complexity of this study. This method creates the opportunity to triangulate and integrate quantitative and qualitative data resulting in a complete and nuanced understanding of complex phenomena . Several strategies are used to enhance the internal validity of the quantitative part. At first, all questionnaires that will be used will be validated and selected after thorough consideration of several researchers with experience in mixed methods implementation research. Secondly, using a wide range of outcome indicators, increases the ability to distinguish confounding from independent variables. Thirdly, if possible a matched controlled group will be used to compare outcomes. Internal validity of qualitative data will be ensured in the stage of data collection by involving researchers who did not participate in the PAR-process to conduct the interviews and focus group interviews. In the stage of data analysis, internal validity of the qualitative data will be enhanced by systematically organizing and coding data and triangulation (data and researcher). Analysis and comparison of the four different settings will reinforce the external validity and transferability of the findings.

ELIGIBILITY:
Patients/parents

Inclusion Criteria:

* Admitted on the participating ward (digestive surgery) or diagnosed stable liver cirrhosis or pediatric epilepsy
* Be conscious
* Speak Dutch

Exclusion Criteria:

- Dementia or other severe cognitive/mental disorders

Health care providers

Inclusion Criteria:

* Have at least three months of clinical experience on the ward
* Key stakeholders in the process of development, implementation and/or evaluation

Exclusion Criteria:

* No contact with the nurse practitioner
* Internship

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients
  - Patients (or their parents in the paediatric department)
  HCPs
  * Representatives of all relevant stakeholders (from each department) will be invited to participate (eg. head(s) of the medical department(s), physicians, physicians in training, (head) nurses, care managers, the chief medical officer, specialised nurses, social worker, pharmacist).
  * All HCPs who are currently involved in the care process of the targeted patient population.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in quality of care NPSS - ambulatory | The data will be collected at three points during the study: baseline T0 (before introduction), T1 (6 months after introduction) and T2 (1 year after introduction)
  Satisfaction with NP/doctor consultation. The data will be collected by use of a questionnaire for patients (and their parents). Validated tools, the Nurse Practitioner Satisfaction Survey (NPSS) and the Quality of care through the patients eyes will be used.
Change in quality of care though the patients eyes - ambulatory liver cirrhosis | The data will be collected at three points during the study: baseline T0 (before introduction), T1 (6 months after introduction) and T2 (1 year after introduction)
  Satisfaction with NP/doctor consultation. The data will be collected by use of a questionnaire for patients (and their parents). A validated tool, the Quality of care through the patients eyes will be used.
Change in Quality of care (GS-PEQ) - hospitalization | The data will be collected at three points during the study: T0 (before introduction), T1 (6 months after introduction) and T2 (1 year after introduction)
  Patient perception and experiences of quality of care provided during hospitalisation. The data will be collected by use of a questionnaire for patients. A validated tool the Generic Short Patient Experiences Questionnaire will be used.
Change in Quality of care (Picker) - hospitalization | The data will be collected at three points during the study: T0 (before introduction), T1 (6 months after introduction) and T2 (1 year after introduction)
  Patient perception and experiences of quality of care provided during hospitalisation. The data will be collected by use of a questionnaire for patients. A validated tool the Picker Patient Experience Questionnaire will be used.

SECONDARY OUTCOMES:
Change in hospital admissions - ambulatory | All admissions one year before and after introduction will be registered. The data will be collected at three points during the study: baseline T0 (before introduction), T1 (6 months after introduction) and T2 (1 year after introduction)
  Number of hospital admissions for patients in ambulatory care. The data will be collected from the patients medical file.
Length of stay hospital admissions - ambulatory | Length of stay of all admissions 12 months before and 12 months after introduction of the Nurse practitioner will be registered.
  Length of stay in hospital for patients in ambulatory care. The data will be collected from the patients medical file.
Change in readmission - hospitalization | The data will be collected at three points during the study: baseline T0 (before introduction), T1 (6 months after introduction) and T2 (1 year after introduction)
  Readmission within seven days after discharge. The data will be collected from the patients medical file.
Change in mortality rates | The data will be collected at three points during the study: baseline T0 (before introduction), T1 (6 months after introduction) and T2 (1 year after introduction)
  Mortality rates of patients included in the study. The data will be collected from the patients medical file.
Change in pain Scores | The data will be collected at three points during the study: baseline T0 (before introduction), T1 (6 months after introduction) and T2 (1 year after introduction)
  Pain scores during hospitalization of surgical patients. The data will be collected from the patiënts medical file. Data will be registered from admission until dismissal.
Change in completeness of recording profile | The data will be collected at three points during the study: baseline T0 (before introduction), T1 (6 months after introduction) and T2 (1 year after introduction)
  Completeness of recording profile within 24h after admission will be registered. The data will be collected from the patients medical file.
Change in timely resignation letters | The data will be collected at three points during the study: baseline T0 (before introduction), T1 (6 months after introduction) and T2 (1 year after introduction)
  Availability of the resignation letter within 24h after admission will be registered. The data will be collected from the patients medical file.
Change in protocol adherence | The data will be collected at three points during the study: baseline T0 (before introduction), T1 (6 months after introduction) and T2 (1 year after introduction)
  Care provided after surgery will be compared to the ERAS-protocol. The data will be collected from the patients medical file.
Change in psychosocial conditions in workplaces | The data will be collected at three points during the study: baseline T0 (before introduction), T1 (6 months after introduction) and T2 (1 year after introduction)
  Psychosocial conditions in workplaces of healthcare providers. The data will be collected by use of a questionnaire for healthcare providers. A validated tool, the Copenhagen Psychosocial Questionnaire (COPSOQ III) will be used.
Change in team collaboration | The data will be collected at three points during the study: baseline T0 (before introduction), T1 (6 months after introduction) and T2 (1 year after introduction)
  Team effectiveness experienced by healthcare providers. The data will be collected by use of a questionnaire for healtcare providers. A validated tool, the Perceptions of Team Effectiveness (PTE) will be used.
Change in effectiveness of mentoring | The data will be collected at three points during the study: T1 (6 months after introduction) and T2 (1 year after introduction)
  Effectiveness of mentoring experienced by the Nurse practitioner and mentor of the Nurse practitioner. The data will be collected by use of individual interviews (mentor and trainee). Additionally data will be collected by use of a questionnaire for trainees. A validated tool, the mentorship effectiveness scale will be used.
Number of medication prescriptions | The data will be collected at three points during the study: baseline T0 (before introduction), T1 (6 months after introduction) and T2 (1 year after introduction)
  Medication prescriptions before and after introduction of the nurse practitioner. The data will be collected from the patients medical file. Data will be registered from admission until dismissal.
Change in selfmanagement liver cirrhosis (HEIQ) | The data will be collected at three points during the study: baseline T0 (before introduction), T1 (6 months after introduction) and T2 (1 year after introduction)
  Knowledge, skills and confidence in selfmanagement. The data will be collected by use of a questionnaire for patients. Avalidated tools, Health Education Impact Questionnaire (HEIQ) for liver cirrhosis will be used.
Change in selfmanagement epilepsy medication (PEMSQ) | The data will be collected at three points during the study: baseline T0 (before introduction), T1 (6 months after introduction) and T2 (1 year after introduction)
  Knowledge, skills and confidence in selfmanagement. The data will be collected by use of a questionnaire for parents of patients. A validated tool, the Pediatric Epilepsy Medication Self-Management Questionnaire (PEMSQ), will be used.
Change in bed occupancy rates | he data will be collected at three points during the study: baseline T0 (before introduction), T1 (6 months after introduction) and T2 (1 year after introduction)
  Bed occupancy rates at the ward before and after introduction of the nurse practitioner. The data will be collected from the administrative files.

OTHER OUTCOMES:
Change in Quality of life (QOL) | The data will be collected at three points during the study: baseline T0 (before introduction), T1 (6 months after introduction) and T2 (1 year after introduction)
  Quality of life in children with epilepsy and patients with liver cirrhosis. The data will be collected by use of a questionnaire for parents of children with epilepsy. Validated tools: the Quality of Life in Childhood Epilepsy Questionnaire (QOLCE-16) Liver disease symptom index and EQ-5D, will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Vermassen, MD, PhD, Principal Investigator — Ghent University/Ghent University Hospital
Locations (2):
- Belgium (2):
  - Ghent University Hospital, Ghent, East Flanders
  - University Hospital Ghent, Ghent

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dehennin L, Kinnaer LM, Vermassen F, Van Hecke A. Role development, implementation and evaluation of nurse practitioners in a Belgian university hospital: a mixed methods study protocol. BMJ Open. 2023 May 3;13(5):e068101. doi: 10.1136/bmjopen-2022-068101. PMID 37137560